CLINICAL TRIAL: NCT04126798
Title: 2BALANCE: the Impact of a Vestibular Dysfunction on Cognitive and Motor Performance in Adults in Single and Dual-task Condition
Brief Title: 2BALANCE: Cognitive-motor Dual-tasking in Persons with Vestibular Disorders
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Universiteit Antwerpen (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: BC-7935
Record Dates: First submitted 2019-02-25; First posted 2019-10-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vestibular Diseases
Keywords: Cognition; Motor performance; Dual-task
MeSH Terms: conditions — Vestibular Diseases | interventions — Memory and Learning Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy adults: Standardization and collecting normative age-related data for cognitive and motor single tasks, as well as cognitive-motor dual-tasks
  Interventions: Other: Behavioural
- Bilateral vestibulopathy: Validation of cognitive and motor single tasks, as well as cognitive-motor dual-tasks
  Interventions: Other: Behavioural
- Unilateral vestibular impairment: Cross-sectional study on cognitive and motor single tasks, as well as cognitive-motor dual-tasks, in persons with unilateral vestibular impairment
  Interventions: Other: Behavioural

INTERVENTIONS:
Other: Behavioural — Assessment of the 2BALANCE protocol: dual-task protocol consisting of a motor task, cognitive task, and motor-cognitive dual-tasks

SUMMARY:
The overall aim of this study is to elucidate the impact of a vestibular dysfunction on the cognitive and motor performance by means of an extensive test protocol, evaluating the vestibular, cognitive and motor function using single as well as dual-task paradigms.

DETAILED DESCRIPTION:
The test protocol consists of five cognitive tasks, all assessing a different cognitive domain: executive function, working memory, processing speed, and visuospatial abilities (mental rotation and visuospatial memory). These cognitive tasks will be performed separately (in single task condition, while seated), as well as while performing different motor tasks (in dual-task condition). These motor tasks will also be performed in single task condition (without performing the cognitive tasks).

The study consists of the establishment of normative age-related data for the single as well as dual-task protocol in healthy adults, age ranging from 18 to 65 years old (objective 1). Subsequently, the test protocol will be validated in persons with bilateral vestibulopathy (objective 2). Finally, a cross-sectional study in persons with unilateral vestibular impairment will take place, and the results on the single as well as dual-task components will be compared to normative data, as well as to persons with bilateral vestibulopathy (objective 3).

ELIGIBILITY:
For healthy controls:

Exclusion Criteria:

* Vestibular disorders or subjective dizziness complains (past or present)
* Hearing loss
* Mild Cognitive Impairment (Montreal Cognitive Assessment, MOCA)
* Visual impairment (Snellen Chart)
* Motor abnormalities (anamnestic questionnaire)

For bilateral vestibulopathy (BV):

Inclusion criteria:

* Bilaterally reduced vestibular function, as defined by the Bárány Criteria for BV(Michael Strupp 2017):
* the horizontal vestibulo-ocular reflex (VOR) gain should be <0.6 bilaterally and/or
* the sum of the maximal peak velocities of caloric response for stimulation with warm and cold water should be <6◦/s bilaterally and/or
* the horizontal angular VOR gain should be <0.1 upon sinusoidal stimulation on the rotation test

For unilateral vestibulopathy:

Inclusion criteria:

* the horizontal VOR gain should be <0.6 unilaterally and/or
* the slow component velocity of the caloric response should be below the age-dependent normative data unilaterally, established by Maes et al. (2010)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults were used for establishing normative data of the dual-task protocol (convenience sampling).
  Persons with bilateral vestibulopathy, established by vestibular assessment, were used for the validation of the study (recruited at the Ghent University Hospital, Antwerp University Hospital, and Maastricht University Medical Center).
  Persons with unilateral vestibular impairment, established by vestibular assessment, were used for the cross-sectional study (recruited at the Ghent University Hospital).
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Stride length measured on the GAITRite Walkway (ProCare) | 4 years
  Stride length measured in centimeters on pressure sensitive mat
Step length measured on the GAITRite Walkway (ProCare) | 4 years
  Step length measured in centimeters on pressure sensitive mat
Stride width measured on the GAITRite Walkway (ProCare) | 4 years
  Stride width measured in centimeters on pressure sensitive mat
Step width measured on the GAITRite Walkway (ProCare) | 4 years
  Step width measured in centimeters on pressure sensitive mat
Step time measured on the GAITRite Walkway (ProCare) | 4 years
  Step time measured in seconds on pressure sensitive mat
Stride time measured on the GAITRite Walkway (ProCare) | 4 years
  Stride time measured in seconds on pressure sensitive mat
Velocity measured on the GAITRite Walkway (ProCare) | 4 years
  Velocity measured in centimeters per second on pressure sensitive mat
Surface (mm²) of the confidence ellipse which contains 90% of the center of pressure (COP) measured on the GymPlate (TechnoConcepts) | 4 years
  Confidence ellipse measured in millimeter² on force platform
Length covered by the consecutive center of pressure (COP) positions measured on the GymPlate (TechnoConcepts) | 4 years
  Length of the COP measured in millimeter on force platform
Mean velocity of the oscillations of the center of pressure (COP) measured on the GymPlate (TechnoConcepts) | 4 years
  Length of the COP measured in millimeter per second on force platform
Velocity variance measured on the GymPlate (TechnoConcepts) | 4 years
  Length of the COP measured in millimeter² per second² on force platform
Percent accuracy on the Corsi Block Test | 4 years
  Measure of visuospatial memory
Response time on the Corsi Block Test | 4 years
  Measure of visuospatial memory in milliseconds
Percentage of accuracy on the mental rotation task | 4 years
  Measure of mental rotation (visuospatial cognition)
Response time on the mental rotation task | 4 years
  Measure of mental rotation (visuospatial cognition) in milliseconds
Percentage of accuracy on the backward digit recall test | 4 years
  Measure of working memory
Response time on the backward digit recall test | 4 years
  Measure of working memory in milliseconds
Percentage of accuracy on the symbol digit modalities test | 4 years
  Measure of processing speed
Response time on the symbol digit modalities test | 4 years
  Measure of processing speed in milliseconds
Percentage of accuracy on the auditory Stroop task | 4 years
  Measure of response inhibition
Response time on the auditory Stroop task | 4 years
  Measure of response inhibition
Percentage of accuracy on the visual Stroop task | 4 years
  Measure of response inhibition
Response time on the visual Stroop task | 4 years
  Measure of response inhibition

CONTACTS AND LOCATIONS:
Overall Officials: Leen Maes, PhD, Principal Investigator — Ghent University Hospital, Ghent University
Locations (1):
- University Hospital Ghent, departement otorhinolaryngology, Ghent, Belgium

REFERENCES:
- [Derived] Danneels M, Van Hecke R, Leyssens L, Degeest S, Cambier D, van de Berg R, Van Rompaey V, Maes L. 2BALANCE: a cognitive-motor dual-task protocol for individuals with vestibular dysfunction. BMJ Open. 2020 Jul 14;10(7):e037138. doi: 10.1136/bmjopen-2020-037138. PMID 32665391